CLINICAL TRIAL: NCT06370975
Title: Effect of 3% Hypertonic Saline Resuscitation on Lactate and Its Comparison With Ringer's Lactated Solution and 0.9% Normal Saline in Traumatic Injury Patients: A Prospective Randomized Control Trial
Brief Title: Effect of Fluid Resuscitation on Lactate in Traumatic Injury Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hevzy Mohamed Ibrahem, DR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fluid resuscitation in trauma
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Fluid Resuscitation
MeSH Terms: interventions — Saline Solution, Hypertonic; Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3% hypertonic Saline (Experimental)
  Interventions: Drug: 3% hypertonic Saline
- Ringer's lactated solution (Experimental)
  Interventions: Drug: Ringer's lactated solution
- 0.9% Normal saline (Experimental)
  Interventions: Drug: 0.9% Normal saline

INTERVENTIONS:
Drug: 3% hypertonic Saline — the patients received 3% HS at the rate of 4 mL/kg for 30 minutes. the intervention period for the study ran for the first hour of treatment, and serial monitoring and lab tests were done during this period, measurement lactate levels will done at 0, 30, 60 mins and 24 hour, the ABG parameters were recorded 30 and 60 min after the completion of the calculated dose infused with fluids and serial monitoring of vital parameters was done at 0, 15, 30, and 60 mins. The lactate clearance was calculated as follows:
  -hour lactate clearance (%) = (0-hour lactate - 1-hour lactate) / 0-hour lactate × 100
  Arms: 3% hypertonic Saline
Drug: Ringer's lactated solution — the patients received ringer's lactated solution at the rate of 20 ml/kg for 30 minute. the intervention period for the study ran for the first hour of treatment, and serial monitoring and lab tests were done during this period, measurement lactate levels will done at 0, 30, 60 mins and 24 hour, the ABG parameters were recorded 30 and 60 min after the completion of the calculated dose infused with fluids and serial monitoring of vital parameters was done at 0, 15, 30, and 60 mins. The lactate clearance was calculated as follows:
  -hour lactate clearance (%) = (0-hour lactate - 1-hour lactate) / 0-hour lactate × 100
  Arms: Ringer's lactated solution
Drug: 0.9% Normal saline — the patients received 0.9% Ns at the rate of 20 ml/kg for 30 minute. the intervention period for the study ran for the first hour of treatment, and serial monitoring and lab tests were done during this period, measurement lactate levels will done at 0, 30, 60 mins and 24 hour, the ABG parameters were recorded 30 and 60 min after the completion of the calculated dose infused with fluids and serial monitoring of vital parameters was done at 0, 15, 30, and 60 mins. The lactate clearance was calculated as follows:
  -hour lactate clearance (%) = (0-hour lactate - 1-hour lactate) / 0-hour lactate × 100
  Arms: 0.9% Normal saline

SUMMARY:
The study aims to investigate the effect of 3% hypertonic saline resuscitation on lactate clearance in comparison to ringer's lactated solution and 0.9% normal saline in traumatic injury patients.

Also to provide insights into the optimal fluid resuscitation strategy for traumatic injury patients

DETAILED DESCRIPTION:
Traumatic injuries considered as important leading causes of morbidity and mortality worldwide; haemorrhagic shock is a common and critical complication. Fluid resuscitation is a crucial step in managing traumatic injury patients, and the choice of resuscitation fluid can significantly impact patient outcomes. In the context of trauma, rapid and effective resuscitation is essential to prevent irreversible cellular dysfunction and multi-organ failure.

Lactate is a key indicator of tissue perfusion and oxygenation in trauma patients, with faster clearance rates associated with improved outcomes. There is growing interest in the use of hypertonic saline for resuscitation in traumatic injury patients, as it may lead to faster lactate clearance compared to traditional crystalloid solutions such as ringer's lactated solution and 0.9% normal saline. Additionally, it has been suggested that hypertonic saline may improve microvascular blood flow and tissue oxygenation, which can aid in lactate clearance. Ringer's lactated solution is commonly used for fluid resuscitation in trauma patients, providing volume expansion and buffering capacity. Furthermore, 0.9% normal saline is widely utilized in clinical practice, but concerns regarding its potential to induce hyperchloremic acidosis have been raised. Given the varied physiological effects of these resuscitative fluids, it is imperative to conduct a robust randomized controlled trial to elucidate their respective impacts on lactate clearance and overall outcomes in traumatic injury patients. Such a comprehensive trial will facilitate evidence-based decision-making and potentially optimize resuscitation strategies in the acute care of trauma patients, ultimately improving survival and reducing the burden of trauma-related morbidity and mortality. To our knowledge there is few studies discussing the differences between the use of 3% hypertonic, ringer's lactated and 0.9% normal salines in urgent resuscitation of trauma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with traumatic injury (e.g., blunt or penetrating trauma, road accidents and patients posted for emergency orthopedic and abdominal surgeries.

2. Patients' ≥ 18 years old.

Exclusion Criteria:

1. Patients with traumatic brain injury or spinal cord injury. 2. Patients with known hypersensitivity or allergy 3% hypertonic, ringer's lactated and 0.9% normal salines.

3. Patients with comorbidities (e.g. pre-existing renal dysfunction, end-stage renal disease, sever liver dysfunction or cirrhosis and coagulopathy or bleeding disorders.

4. Patients with serum electrolyte abnormalities who required inotropic support at the time of presentation.

5. Patients who are pregnant or burns trauma. 6. Patients receiving concurrent treatment with hypertonic solutions for other conditions.

7. Patients refused to participate or continuation in the study. 8. Deaths directly due to trauma were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Rate of lactate clearance following resuscitation with different solutions | baseline
  assess lactate clearance in traumatic patients after resuscitation with 3% hypertonic saline, ringer's lactated saline and 0.9% normal saline